CLINICAL TRIAL: NCT05459038
Title: Clinical Validation of the C-Arm Rotational View (CARV) to Avoid Rotational Malalignment After Intramedullary Nailing of Tibial Shaft Fractures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 81191
Record Dates: First submitted 2022-04-05; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Tibial Fractures; Surgery; Complication,Postoperative
Keywords: Intramedullary nailing; Tibia shaft fractures; Rotational malalignment; C-Arm Rotational View; multi-center randomized controlled trial.
MeSH Terms: conditions — Tibial Fractures; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Multi-center randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Patients assigned to the interventional group will undergo an identical surgical procedure as patients assigned to the control group. The only difference with the control group is that tibial alignment will be obtained according to the standardized CARV-protocol.
  Interventions: Diagnostic Test: C-Arm Rotational View (CARV)
- Control group (No Intervention): Patients assigned to the control group will undergo an identical surgical procedure as patients assigned to the interventional group. The only difference with the intervention group is that tibial alignment will be obtained according to present unstandardized clinical standards

INTERVENTIONS:
Diagnostic Test: C-Arm Rotational View (CARV) — CARV includes predefined fluoroscopy landmarks of the uninjured side to correct for rotational malalignment of the injured side in which the rotation of the C-Arm Image Intensifier is used
  Arms: Interventional group

SUMMARY:
Tibia shaft fractures are common long bone fractures in the field of Orthopaedic Trauma. In the USA, a total of 492.000 tibial fractures were reported per year by the National Center of Health Statistics (NCHS). Intramedullary nailing (IMN) is the treatment of choice for shaft fractures. However, rotational malalignment (RM) remains an iatrogenic pitfall with a prevalence up to 30%.

From a clinical point of view, there is limited knowledge on how to avoid RM during IMN. Clinical estimation of tibial alignment is difficult, resulting frequently in RM following IMN. Low-dose CT-assessment is considered the gold standard to objectify RM, but is performed after surgery when the opportunity for direct revision has passed. Both difficulties in intraoperative clinical judgement of tibial alignment as well as postoperative detection of RM when the possibility for direct revision has passed, do support the need for an easy-to-use intraoperative fluoroscopy protocol to minimize the risk for RM during IMN of tibial shaft fractures.

Recently, a standardized intraoperative fluoroscopy protocol named the 'C-Arm Rotational View (CARV)' was determined in order to improve the accuracy of alignment control during IMN of tibial shaft fractures. CARV includes predefined fluoroscopy landmarks of the uninjured side to correct for rotational malalignment of the injured side in which the rotation of the C-Arm Image Intensifier is used. Promising preliminary results were found to reduce the risk on RM following IMN of tibia fractures. However, a prospective trial is needed to determine the performance of CARV in clinical practice. Therefore, a prospective multi-center randomized controlled trial is designed to assess the clinical feasibility and potential benefits of the CARV-protocol. The following primary research question was defined: can the risk for RM following IMN of tibial shaft fractures be minimized by use of the CARV-protocol?

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients (≥18 years) with an open or closed tibia shaft fracture, who are eligible for IMN, will be asked to enroll in the study

Exclusion Criteria:

* The following exclusion criteria will be used: age <18 years, fractures not suitable for IMN and pathological fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rotational (mal)alignment | Up to 12 months after initial surgery
  Determine the incidence of RM using postoperative CT-assessment. In literature, RM is defined as a rotation ≥10 degrees relative to the contralateral side. However, considering the physiological left-right difference of 4 degrees between left and right-sided tibiae, with right-sided tibiae on average 4 degrees more externally rotated, RM is defined as malrotation of < -6 degrees or >14 degrees in right-sided tibiae and < -14 degrees or >6 degrees in left-sided tibiae. A negative angle represents internal rotation and positive angle external rotation.

CONTACTS AND LOCATIONS:
Locations (2):
- Flinders Medical Centre, Flinders University, Adelaide, Australia
- University Medical Centers Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Theriault B, Turgeon AF, Pelet S. Functional impact of tibial malrotation following intramedullary nailing of tibial shaft fractures. J Bone Joint Surg Am. 2012 Nov 21;94(22):2033-9. doi: 10.2106/JBJS.K.00859. PMID 23172320
- [Background] Cain ME, Hendrickx LAM, Bleeker NJ, Lambers KTA, Doornberg JN, Jaarsma RL. Prevalence of Rotational Malalignment After Intramedullary Nailing of Tibial Shaft Fractures: Can We Reliably Use the Contralateral Uninjured Side as the Reference Standard? J Bone Joint Surg Am. 2020 Apr 1;102(7):582-591. doi: 10.2106/JBJS.19.00731. PMID 31977824
- [Background] Bleeker NJ, Cain M, Rego M, Saarig A, Chan A, Sierevelt I, Doornberg JN, Jaarsma RL. Bilateral Low-Dose Computed Tomography Assessment for Post-Operative Rotational Malalignment After Intramedullary Nailing for Tibial Shaft Fractures: Reliability of a Practical Imaging Technique. Injury. 2018 Oct;49(10):1895-1900. doi: 10.1016/j.injury.2018.07.031. Epub 2018 Jul 29. PMID 30097311
- [Background] Puloski S, Romano C, Buckley R, Powell J. Rotational malalignment of the tibia following reamed intramedullary nail fixation. J Orthop Trauma. 2004 Aug;18(7):397-402. doi: 10.1097/00005131-200408000-00001. PMID 15289683
- [Background] Bleeker NJ, Reininga IHF, van de Wall BJM, Hendrickx LAM, Beeres FJP, Duis KT, Doornberg JN, Jaarsma RL, Kerkhoffs GMMJ, IJpma FFA. Difference in Pain, Complication Rates, and Clinical Outcomes After Suprapatellar Versus Infrapatellar Nailing for Tibia Fractures? A Systematic Review of 1447 Patients. J Orthop Trauma. 2021 Aug 1;35(8):391-400. doi: 10.1097/BOT.0000000000002043. PMID 34267147
- [Background] Shih YC, Chau MM, Arendt EA, Novacheck TF. Measuring Lower Extremity Rotational Alignment: A Review of Methods and Case Studies of Clinical Applications. J Bone Joint Surg Am. 2020 Feb 19;102(4):343-356. doi: 10.2106/JBJS.18.01115. No abstract available. PMID 31743239
- [Derived] Bleeker NJ, Doornberg JN, Ten Duis K, El Moumni M, Jaarsma RL, IJpma FFA. Clinical validation of the 'C-arm rotational view (CARV)': study protocol of a prospective randomised controlled trial. BMJ Open. 2023 Nov 22;13(11):e064802. doi: 10.1136/bmjopen-2022-064802. PMID 37993156